CLINICAL TRIAL: NCT04342494
Title: Providing Mental Health Precision Treatment
Acronym: PROMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amy S.B. Bohnert, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00164162
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Depression; Addiction; Anxiety; Sleep Disturbance
Keywords: Behavioral health; Precision health
MeSH Terms: conditions — Depression; Behavior, Addictive; Anxiety Disorders; Parasomnias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (5):
- Enhanced Feedback + Standard Feedback (Experimental): Participants will receive enhanced feedback from the MyDataHelps study app in addition to standard feedback from the activity tracker.
  Interventions: Behavioral: Enhanced Feedback + Standard Feedback
- Headspace app + Standard Feedback (Experimental): Participants will receive an app-based intervention in addition to standard feedback from the activity tracker.
  Interventions: Device: Headspace app + Standard Feedback
- Headspace app + Enhanced Feedback + Standard Feedback (Experimental): Participants will receive an app-based intervention, enhanced feedback from the MyDataHelps study app, and standard feedback activity tracker.
  Interventions: Device: Headspace app + Enhanced Feedback + Standard Feedback
- SilverCloud app + Standard Feedback (Experimental): Participants will receive an app-based intervention in addition to standard feedback from the activity tracker.
  Interventions: Device: SilverCloud + Standard Feedback
- SilverCloud app +Enhanced Feedback +Standard Feedback (Experimental): Participants will receive an app-based intervention, enhanced feedback from the MyDataHelps study app, and standard feedback from the activity tracker.
  Interventions: Device: SilverCloud app +Enhanced Feedback +Standard Feedback

INTERVENTIONS:
Behavioral: Enhanced Feedback + Standard Feedback — Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Enhanced Feedback (EF) Participants randomized to receive enhanced feedback will receive this feedback from the MyDataHelps study app. This includes varying types of text and visual feedback based on data collected through the app. Feedback will be displayed to participants on a dashboard in the app or delivered via pop-up notifications. Participants will receive a combination of text and visual feedback.
  Arms: Enhanced Feedback + Standard Feedback
Device: Headspace app + Standard Feedback — Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Headspace is an app designed to train the user in mindfulness practices.
  Arms: Headspace app + Standard Feedback
Device: Headspace app + Enhanced Feedback + Standard Feedback — Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Enhanced Feedback (EF) Participants randomized to receive enhanced feedback will receive this feedback from the MyDataHelps study app. This includes varying types of text and visual feedback based on data collected through the app. Feedback will be displayed to participants on a dashboard in the app or delivered via pop-up notifications. Participants will receive a combination of text and visual feedback.
  Headspace is an app designed to train the user in mindfulness practices.
  Arms: Headspace app + Enhanced Feedback + Standard Feedback
Device: SilverCloud + Standard Feedback — Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Silvercloud is an app designed to deliver cognitive behavioral therapy.
  Arms: SilverCloud app + Standard Feedback
Device: SilverCloud app +Enhanced Feedback +Standard Feedback — Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Enhanced Feedback (EF) Participants randomized to receive enhanced feedback will receive this feedback from the MyDataHelps study app. This includes varying types of text and visual feedback based on data collected through the app. Feedback will be displayed to participants on a dashboard in the app or delivered via pop-up notifications. Participants will receive a combination of text and visual feedback.
  Silvercloud is an app designed to deliver cognitive behavioral therapy.
  Arms: SilverCloud app +Enhanced Feedback +Standard Feedback

SUMMARY:
This research study is being conducted to understand if patients benefit from mobile health interventions while waiting for in-clinic mental health treatments, and to understand which patients receive the most benefit.

DETAILED DESCRIPTION:
Initially, results-reporting was planned for 12-month data. However, following 6-week data collection, the participants received other care, so the decision was made to report on the 6-week data.

ELIGIBILITY:
Inclusion Criteria:

* Must have a scheduled mental health intake appointment at Michigan Medicine Outpatient Psychiatry or University Health Service at the University of Michigan
* Must have daily access to a smartphone version that is compatible with study activity trackers.
* Understands English to enable consent and use of the MyDataHelps app and app-based interventions
* Provide complete, updated contact information upon enrollment to the study
* Agree to be contacted by study staff during the study
* Willingness to keep study setup (devices, apps, settings) in required configuration for the duration of the study, and following instructions by study staff if required to update or re-achieve required configuration if required configuration has been lost (e.g., change of phone, app deletion)

Exclusion Criteria:

* Self-reported or medical record indication of a current eating disorder
* Scheduled outpatient mental health appointment is a pediatric appointment (even if age 18+)
* Wrist too large or too small to wear an Apple Watch or Fitbit comfortably (Note: bands that are shorter or longer than the standard will be made available to minimize this exclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2118 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Bohnert, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horwitz AG, Mills ED, Sen S, Bohnert ASB. Comparative Effectiveness of Three Digital Interventions for Adults Seeking Psychiatric Services: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2422115. doi: 10.1001/jamanetworkopen.2024.22115. PMID 39023893

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2118 participants were consented for this trial. Of that number, 2079 completed baseline and were randomized.
Groups:
- Enhanced Feedback + Standard Feedback: Participants will receive enhanced feedback from the MyDataHelps study app in addition to standard feedback from the activity tracker.
  Enhanced Feedback + Standard Feedback: Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Enhanced Feedback (EF) Participants randomized to receive enhanced feedback will receive this feedback from the MyDataHelps study app. This includes varying types of text and visual feedback based on data collected through the app. Feedback will be displayed to participants on a dashboard in the app or delivered via pop-up notifications. Participants will receive a combination of text and visual feedback.
- Headspace App + Standard Feedback: Participants will receive an app-based intervention in addition to standard feedback from the activity tracker.
  Headspace app + Standard Feedback: Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Headspace is an app designed to train the user in mindfulness practices.
- Headspace App + Enhanced Feedback + Standard Feedback: Participants will receive an app-based intervention, enhanced feedback from the MyDataHelps study app, and standard feedback activity tracker.
  Headspace app + Enhanced Feedback + Standard Feedback: Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Enhanced Feedback (EF) Participants randomized to receive enhanced feedback will receive this feedback from the MyDataHelps study app. This includes varying types of text and visual feedback based on data collected through the app. Feedback will be displayed to participants on a dashboard in the app or delivered via pop-up notifications. Participants will receive a combination of text and visual feedback.
  Headspace is an app designed to train the user in mindfulness practices.
- SilverCloud App + Standard Feedback: Participants will receive an app-based intervention in addition to standard feedback from the activity tracker.
  SilverCloud + Standard Feedback: Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Silvercloud is an app designed to deliver cognitive behavioral therapy.
- SilverCloud App +Enhanced Feedback +Standard Feedback: Participants will receive an app-based intervention, enhanced feedback from the MyDataHelps study app, and standard feedback from the activity tracker.
  SilverCloud app +Enhanced Feedback +Standard Feedback: Standard Feedback (SF) All participants will receive the standard feedback that is standard feedback from the activity trackers. Feedback includes activity level, heart rate, and progress toward daily activity goals on the device itself.
  Enhanced Feedback (EF) Participants randomized to receive enhanced feedback will receive this feedback from the MyDataHelps study app. This includes varying types of text and visual feedback based on data collected through the app. Feedback will be displayed to participants on a dashboard in the app or delivered via pop-up notifications. Participants will receive a combination of text and visual feedback.
  Silvercloud is an app designed to deliver cognitive behavioral therapy.
Period: Overall Study
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback
Started | 690 | 349 | 349 | 345 | 346
Completed | 640 | 311 | 313 | 311 | 310
Not Completed | 50 | 38 | 36 | 34 | 36
Not completed — Questionnaire partially completed | 1 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 49 | 38 | 34 | 34 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback | Total
Number analyzed (Participants) | 690 | 349 | 349 | 345 | 346 | 2079
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (14.5) | 36.2 (14.4) | 36.8 (14.5) | 36.8 (13.7) | 36.5 (14.3) | 36.8 (14.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 192 | 80 | 106 | 89 | 93 | 560
  Female | 491 | 267 | 242 | 251 | 248 | 1499
  Unknown | 7 | 2 | 1 | 5 | 5 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 28 | 31 | 24 | 15 | 142
  Not Hispanic or Latino | 641 | 318 | 314 | 319 | 328 | 1920
  Unknown or Not Reported | 5 | 3 | 4 | 2 | 3 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 1 | 2 | 8
  Asian | 44 | 17 | 17 | 17 | 23 | 118
  Black | 57 | 33 | 23 | 31 | 18 | 162
  White | 516 | 269 | 275 | 259 | 271 | 1590
  Multiple races | 38 | 12 | 16 | 17 | 16 | 99
  Other | 27 | 13 | 11 | 16 | 11 | 78
  Unknown | 6 | 4 | 5 | 4 | 5 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 690 | 349 | 349 | 345 | 346 | 2079
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 495 | 241 | 253 | 236 | 223 | 1448
  Bisexual | 91 | 53 | 44 | 50 | 63 | 301
  Gay or lesbian | 29 | 14 | 18 | 27 | 17 | 105
  Other | 35 | 24 | 13 | 16 | 22 | 110
  Multiple identities | 20 | 8 | 10 | 8 | 10 | 56
  Unknown | 20 | 9 | 11 | 8 | 11 | 59
Employment Status [Count of Participants; unit: Participants]
  Full-time | 261 | 136 | 150 | 141 | 137 | 825
  Part-time | 140 | 61 | 61 | 66 | 71 | 399
  Retired | 53 | 24 | 21 | 20 | 21 | 139
  Student | 91 | 53 | 42 | 45 | 47 | 278
  Unemployed | 143 | 75 | 75 | 72 | 70 | 435
  Unknown | 2 | 0 | 0 | 1 | 1 | 4
Educational Level [Count of Participants; unit: Participants]
  <High school diploma | 14 | 7 | 12 | 6 | 9 | 48
  High school diploma or GED | 68 | 38 | 37 | 44 | 38 | 225
  Some College | 165 | 98 | 85 | 86 | 85 | 519
  Associate degree or TVS | 88 | 45 | 52 | 37 | 39 | 261
  Bachelor's degree | 207 | 84 | 95 | 84 | 94 | 564
  ≥Master's degree | 146 | 77 | 68 | 87 | 80 | 458
  Unknown | 2 | 0 | 0 | 1 | 1 | 4
Gender Identity [Count of Participants; unit: Participants]
  Man | 192 | 78 | 97 | 84 | 88 | 539
  Woman | 466 | 248 | 231 | 242 | 236 | 1423
  Transgender and Nonbinary (TGNB) | 28 | 19 | 21 | 18 | 20 | 106
  Unknown | 4 | 4 | 0 | 1 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression as Measured by the Patient Health Questionnaire 9 (PHQ-9)
Description: The PHQ-9 was a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 incorporated self-report questions on 9 specific depression symptoms that align with the DSM-IV depression diagnostic criteria. PHQ-9 scores ranged from 0-27, with 0 indicating no depression and 27 indicating severe depression.
Time Frame: Up to 6 weeks
Population: Some participants in each arm were lost to follow up or did not complete their questionnaires following the baseline visit. 1 participant's data for the PHQ-9 was missing, but their data for Outcome Measures 3, 4, 5, and 6 was present.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback
Number analyzed (Participants) | 690 | 349 | 349 | 345 | 346
score on a scale
  Baseline | 12.6 (6.4) | 12.5 (6.3) | 13.0 (6.8) | 13.0 (6.2) | 12.8 (6.4)
  6 weeks: number analyzed (Participants) | 640 | 311 | 313 | 311 | 310
  6 weeks | 10.1 (5.8) | 9.8 (5.9) | 10.1 (5.9) | 10.3 (5.9) | 10.6 (5.7)
Statistical Analysis 1: Comparison: Enhanced Feedback + Standard Feedback vs Headspace App + Standard Feedback vs Headspace App + Enhanced Feedback + Standard Feedback vs SilverCloud App + Standard Feedback vs SilverCloud App +Enhanced Feedback +Standard Feedback; Test type: Equivalence — Symptom-level change estimates were adjusted for baseline PHQ-9 score via analysis of covariance; p = 0.31, ANCOVA

2. Secondary Outcome: Mood as Measured by the Mental Health App Assessment
Description: Participants were asked a single question, "On a scale of 1 to 10, what was your average mood today?" Scores were averaged over follow-up periods with lower scores indicating worse moods and higher scores indicating better moods.
Time Frame: Daily up to 6 weeks
Population: Only participants who completed their mood scores between weeks 2 and 6 were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback
Number analyzed (Participants) | 681 | 346 | 344 | 340 | 341
score on a scale | 6.2 (1.4) | 6.1 (1.3) | 6.2 (1.4) | 6.0 (1.3) | 5.9 (1.4)
Statistical Analysis 1: Comparison: Enhanced Feedback + Standard Feedback vs Headspace App + Standard Feedback vs Headspace App + Enhanced Feedback + Standard Feedback vs SilverCloud App + Standard Feedback vs SilverCloud App +Enhanced Feedback +Standard Feedback; Test type: Equivalence — Average mood score obtained from daily measurements analyzed via analysis of variance; p = 0.0073, ANOVA

3. Secondary Outcome: Change in Suicide Risk as Measured by the Positive and Negative Suicide Ideation Inventory - Positive Ideation (PANSI-PI)
Description: The PANSI-PI subscale consisted of 6 items. The possible total scores on the PANSI-PI subscale ranged from 6 to 30. Lower scores on the PANSI-PI reflected greater risk for suicidal behavior.
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback
Number analyzed (Participants) | 690 | 349 | 349 | 345 | 346
score on a scale
  Baseline | 18.4 (5.0) | 18.4 (5.1) | 17.9 (5.1) | 18.2 (4.9) | 17.8 (5.3)
  6 weeks: number analyzed (Participants) | 641 | 311 | 313 | 311 | 310
  6 weeks | 19.1 (5.3) | 19.6 (5.6) | 19.0 (5.1) | 18.8 (4.9) | 18.2 (5.3)
Statistical Analysis 1: Comparison: Enhanced Feedback + Standard Feedback vs Headspace App + Standard Feedback vs Headspace App + Enhanced Feedback + Standard Feedback vs SilverCloud App + Standard Feedback vs SilverCloud App +Enhanced Feedback +Standard Feedback; Test type: Equivalence — Symptom-level change estimates were adjusted for baseline PANSI-PI score via analysis of covariance; p = 0.03, ANCOVA

4. Secondary Outcome: Change in Suicide Risk as Measured by the Positive and Negative Suicide Ideation Inventory - Negative Suicide Ideation (PANSI-NSI)
Description: The PANSI-NSI subscale was composed of 8 items. The possible total score on the PANSI-NSI ranged from 8 to 40. Higher scores on the PANSI-NSI reflected greater risk for suicidal behavior.
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback
Number analyzed (Participants) | 690 | 349 | 349 | 345 | 346
score on a scale
  Baseline | 11.1 (5.8) | 11.0 (5.6) | 12.2 (6.8) | 11.6 (6.8) | 11.7 (6.3)
  6 weeks: number analyzed (Participants) | 641 | 311 | 313 | 311 | 310
  6 weeks | 9.9 (4.6) | 9.9 (4.4) | 10.8 (5.5) | 10.5 (5.5) | 10.6 (5.0)
Statistical Analysis 1: Comparison: Enhanced Feedback + Standard Feedback vs Headspace App + Standard Feedback vs Headspace App + Enhanced Feedback + Standard Feedback vs SilverCloud App + Standard Feedback vs SilverCloud App +Enhanced Feedback +Standard Feedback; Test type: Equivalence — Symptom-level change estimates were adjusted for baseline PANSI-NSI score via analysis of covariance; p = 0.71, ANCOVA

5. Secondary Outcome: Change in Anxiety as Measured Using the Generalized Anxiety Disorder 7-Item (GAD-7) Scale
Description: GAD-7 consisted of the total score for seven items ranging from 0 to 21. Scores of 5, 10, and 15 represented cut points for mild, moderate, and severe anxiety, respectively.
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback
Number analyzed (Participants) | 690 | 349 | 349 | 345 | 346
score on a scale
  Baseline | 11.5 (5.8) | 11.6 (5.8) | 11.4 (5.9) | 11.9 (6.0) | 11.8 (5.8)
  6 weeks: number analyzed (Participants) | 641 | 311 | 313 | 311 | 311
  6 weeks | 9.9 (5.9) | 9.5 (5.4) | 9.7 (5.7) | 10.0 (5.6) | 9.8 (5.7)
Statistical Analysis 1: Comparison: Enhanced Feedback + Standard Feedback vs Headspace App + Standard Feedback vs Headspace App + Enhanced Feedback + Standard Feedback vs SilverCloud App + Standard Feedback vs SilverCloud App +Enhanced Feedback +Standard Feedback; Test type: Equivalence — Symptom-level change estimates were adjusted for baseline GAD-7 score via analysis of covariance; p = 0.31, ANCOVA

6. Secondary Outcome: Substance Use as Measured by the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST)
Description: The ASSIST Global Continuum of Illicit Drug Risk Score ranged from 0 to 308, with higher scores indicating greater risk. Results reflect the participants who indicated they had consumed any alcohol, smoked, or used an illicit substance when asked.
Time Frame: Up to 6 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback
Number analyzed (Participants) | 690 | 349 | 349 | 345 | 346
Participants
  Baseline | 560 | 300 | 303 | 287 | 285
  6 weeks: number analyzed (Participants) | 641 | 311 | 313 | 311 | 311
  6 weeks | 510 | 253 | 263 | 255 | 247

ADVERSE EVENTS:
Time Frame: Up to 6 weeks
Arm/Group | Enhanced Feedback + Standard Feedback | Headspace App + Standard Feedback | Headspace App + Enhanced Feedback + Standard Feedback | SilverCloud App + Standard Feedback | SilverCloud App +Enhanced Feedback +Standard Feedback
All-Cause Mortality (participants affected / at risk) | 0/690 | 0/349 | 0/349 | 0/345 | 0/346
Serious Adverse Events (participants affected / at risk) | 0/690 | 0/349 | 0/349 | 0/345 | 0/346
Other Adverse Events (participants affected / at risk) | 0/690 | 0/349 | 0/349 | 0/345 | 0/346

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT04342494/Prot_SAP_000.pdf